CLINICAL TRIAL: NCT00586469
Title: Observer-blind, Post-Marketing Study to Compare the Safety and Immunogenicity of Fluviral® Trivalent Split Virion Influenza Vaccine (2007-2008 Season) Made With New vs. Aged Bulk Material, in Adults Ranging in Age From 18 to 60 Years
Brief Title: A Randomized Study to Compare the Safety and Immunogenicity of Fluviral® Made With New Versus Aged Bulk
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 111258
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2009-05-28 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Influenza Vaccines
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Old Bulk (Experimental): This group receives a full dose of Fluviral made from aged bulk material
  Interventions: Biological: Fluviral
- New Bulk (Active Comparator): This group receives a full dose of Fluviral made from new material
  Interventions: Biological: Fluviral

INTERVENTIONS:
Biological: Fluviral — One dose, Intramuscular injection

SUMMARY:
Vaccination is currently the most effective means of controlling influenza and preventing its complications and mortality in persons at risk.

Once a year, a meeting of World Health Organization (WHO) experts takes place, leading to a recommendation on the influenza A and B strains that should be used for the production of vaccine for the coming influenza season. For the strains which do not change from the previous year, the vaccine can be formulated from the old mono bulk from the previous year.

Bulks as old as 12 months may be blended to make trivalent inactivated vaccine (TIV) under the current Canadian and US licenses. This study is conducted to evaluate safety and immunogenicity of Fluviral vaccines made with the aged bulk material compared with the new bulk material. This protocol posting has been updated in order to comply with the FDA Amendment Act, Sept 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol should be enrolled in the study.
* Male and female adults, 18 to 60 years.
* Written informed consent obtained from the subject.
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for the duration of the study.

Exclusion Criteria:

* Acute disease at the time of enrollment.
* Any confirmed or suspected immunosuppressive condition
* Presence of blood dyscrasias, including hemaglobinopathies and myelo- or lymphoproliferative disorder.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* A history of any demyelinating disease including Guillain-Barré syndrome.
* Presence of an active neurological disorder.
* Any significant disorder of coagulation that increases the risk of intramuscular injections or treatment with coumadin derivatives or heparin.
* Receipt of an influenza vaccine within 6 months prior to study enrollment.
* Administration of any vaccines within 30 days prior to study enrollment or during the study period.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the vaccination or planned use during the study period.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or planned during the study.
* Any known or suspected allergy to any constituent of Fluviral and/or a history of anaphylactic type reaction to consumption of eggs, and/or reactions to products containing mercury.
* A history of severe adverse reaction to a previous influenza vaccination.
* Lactating/nursing female.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2007-12-14 (Actual); Primary Completion 2008-01-14 (Actual); Study Completion 2008-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Canada (6):
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 111258 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111258 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111258 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111258 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111258 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111258 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111258 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Old Bulk: This group received a full dose of Fluviral made from aged bulk material
- New Bulk: This group received a full dose of Fluviral made from new material
Period: Overall Study
Arm/Group | Old Bulk | New Bulk
Started | 500 | 500
Completed | 500 | 499
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Old Bulk | New Bulk | Total
Number analyzed (Participants) | 500 | 500 | 1000
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (12.08) | 40.1 (12.01) | 40.1 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 296 | 280 | 576
  Male | 204 | 220 | 424

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Anti-H3 and B Strains
Description: GMTs for H1 strain is addressed as a secondary endpoint
Time Frame: At Day 21
Population: Analysis was performed on the According-To-Protocol cohort for immunogenicity, including subjects for whom results were available for that particular timepoint and who were not eliminated due to exclusion criteria.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Old Bulk | New Bulk
Number analyzed (Participants) | 298 | 291
Titer
  Anti-H3N2 antibody GMT | 369.6 [323.4 to 422.4] | 331.2 [288.8 to 379.7]
  Anti-B antibody GMT | 269.6 [241.6 to 300.9] | 245.0 [216.7 to 276.9]

2. Secondary Outcome: Geometric Mean Titers (GMTs) of the H1 Strain and the GMT of the H3 and B Strains
Description: The table contains GMTs of the H1 strains at Day 0 & 21 and of the H3 and B strains at Day 0 (values at Day 21 for H3 and B strains were primary outcome measures)
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Old Bulk | New Bulk
Number analyzed (Participants) | 298 | 292
Titer
  Anti-H1N1 antibody GMT at Day 0 (n=297, 292) | 15.1 [13.1 to 17.4] | 15.7 [13.6 to 18.1]
  Anti-H1N1 antibody GMT at Day 21 (n=298, 291) | 188.1 [163.6 to 216.4] | 169.9 [147.3 to 196.1]
  Anti-H3N2 antibody GMT at Day 0 (n=297, 292) | 30.4 [25.8 to 35.9] | 35.7 [30.1 to 42.3]
  Anti-B antibody GMT at Day 0 (n=297, 292) | 29.3 [25.3 to 33.9] | 30.0 [25.8 to 34.9]

3. Secondary Outcome: Number of Participants Who Seroconverted.
Description: The table shows the number of participants who have either a pre-vaccination titer < 1:10 and a post-vaccination titer >= 1:40 or a prevaccination titer >= 1:10 and at least a 4-fold increase in post-vaccination titer, at Day 21.
Time Frame: At Day 21.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Old Bulk | New Bulk
Number analyzed (Participants) | 297 | 291
participants
  Anti-H1N1 | 218 | 197
  Anti-H3N2 | 212 | 187
  Anti-B | 205 | 185

4. Secondary Outcome: Number of Seroprotected Participants.
Description: The table presents the number of participants with a serum haemagglutination inhibition (HI) titer >= 1:40 that usually is accepted as indicating protection.
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Old Bulk | New Bulk
Number analyzed (Participants) | 298 | 292
participants
  Anti-H1N1 at Day 0 (n=297, 292) | 80 | 90
  Anti-H1N1 at Day 21 (n=298, 291) | 276 | 266
  Anti-H3N2 at Day 0 (n=297, 292) | 149 | 154
  Anti-H3N2 at Day 21 (n=298, 291) | 293 | 286
  Anti-B antibody GMT at Day 0 (n=297, 292) | 144 | 150
  Anti-B antibody GMT at Day21 (n=298, 291) | 295 | 285

5. Secondary Outcome: Seroconversion Factors Defined as the Fold Increase in Serum HI GMTs Post-vaccination for Influenza Antigen H1N1
Description: Seroconversion factors are defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0, at Day 21. This table presents the SCF for the H1 strain. The SCF for the other strains are addressed in the next table.
Time Frame: At Day 21 compared to Day 0
Population: as for outcome 1
Measure: Number; unit: Factor
Arm/Group | Old Bulk | New Bulk
Number analyzed (Participants) | 297 | 291
Factor | 12.5 | 10.8

6. Secondary Outcome: The Fold Increase in Anti-HI GMTs for Influenza Antigens H3 and B
Description: The fold increase in anti-HI GMTs for influenza antigen H1 is presented in the previous table. The "fold increase" corresponds to the Unit of Measure "Factor."
Time Frame: At Day 21 compared to Day 0
Population: as for outcome 1
Measure: Number; unit: Factor
Arm/Group | Old Bulk | New Bulk
Number analyzed (Participants) | 297 | 291
Factor
  Anti-H3N2 | 12.1 | 9.2
  Anti-B | 9.2 | 8.1

7. Secondary Outcome: Number of Participants Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling.
Time Frame: During the 4-day follow up period following vaccination.
Population: Analysis was performed on the Total Vaccinated cohort.
Measure: Number; unit: participants
Arm/Group | Old Bulk | New Bulk
Number analyzed (Participants) | 500 | 500
participants
  Pain | 271 | 290
  Redness | 88 | 97
  Swelling | 59 | 63

8. Secondary Outcome: Number of Participants Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include bronchospasm, chills, cough, fatigue, fever, headache, joint pain at other location, muscle aches, red eyes, sore throat, and swelling of the face
Time Frame: During the 4-day period following each vaccination.
Population: Analysis was performed on the Total Vaccinated cohort.
Measure: Number; unit: participants
Arm/Group | Old Bulk | New Bulk
Number analyzed (Participants) | 500 | 500
participants
  Bronchospasm | 26 | 24
  Chills | 60 | 45
  Cough | 50 | 53
  Fatigue | 113 | 113
  Axillary fever >= 37.5° Celsius (C) | 18 | 9
  Headache | 110 | 101
  Joint pain at other location | 55 | 50
  Muscle aches | 141 | 138
  Red eyes | 32 | 31
  Sore throat | 61 | 62
  Swelling of the face | 9 | 11

9. Secondary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AE).
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 21-day period following each vaccination.
Population: The analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: participants
Arm/Group | Old Bulk | New Bulk
Number analyzed (Participants) | 500 | 500
participants | 127 | 129

10. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAE)
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: Within 21 days after vaccination
Measure: Number; unit: participants
Arm/Group | Old Bulk | New Bulk
Number analyzed (Participants) | 500 | 500
participants
  Any SAE | 0 | 4
  Fatal SAE | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs were reported during the 4-day follow up period following vaccination; unsolicited AEs during the 21-day period following each vaccination and SAEs during the entire study period (within 21 days after vaccination)
Description: For this study, the Total Number (#) of Participants Affected by Other (non-serious) Adverse Events (AEs) was analyzed separately for expected AEs and for unexpected AEs. A consolidated analysis of all expected and unexpected AEs was not technically possible to be performed and the relevant data are no longer available. Therefore, the Total #Participants Affected in Other Adverse Events Table is currently populated by the highest value of #Participants affected within other AE's table.
Arm/Group | Old Bulk | New Bulk
All-Cause Mortality (participants affected / at risk) | 0/500 | 0/500
Serious Adverse Events (participants affected / at risk) | 0/500 | 4/500
Other Adverse Events (participants affected / at risk) | 271/500 | 290/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Old Bulk (N=500) | New Bulk (N=500)
Drug hypersensitivity (Immune system disorders) | 0 | 2
Bipolar disorder (Psychiatric disorders) | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Old Bulk (N=500) | New Bulk (N=500)
Nasopharyngitis (Infections and infestations) | 19 | 26
Pain (General disorders) | 271 | 290
Redness (General disorders) | 88 | 97
Swelling (General disorders) | 59 | 63
Bronchospasm (General disorders) | 26 | 24
Chills (General disorders) | 60 | 45
Cough (General disorders) | 50 | 53
Fatigue (General disorders) | 113 | 113
Headache (General disorders) | 110 | 101
Joint pain at other location (General disorders) | 55 | 50
Muscle aches (General disorders) | 141 | 138
Red eyes (General disorders) | 32 | 31
Sore throat (General disorders) | 61 | 62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.